CLINICAL TRIAL: NCT03415841
Title: Kardia - A Smartphone-based Care Model for Outpatient Cardiac Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Collaborators: Biofourmis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Kardia
Record Dates: First submitted 2017-10-24; First posted 2018-01-30 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Post MI
Keywords: Post MI; Cardiac Rehabilitation; Wearable Devices; Smartphone-based Program

STUDY DESIGN:
Intervention Model Description: 50 patients who are randomized to the intervention group (mHealth) will be enabled with remote monitoring devices (Blood Pressure and wearable vital signs monitor, Biovotion) and "Kardia" mobile application, for home-based rehabilitation program followed by review in the outpatient Cardiology clinics. The control group (50 patients) will just be monitored at fixed intervals in the outpatient Cardiology clinics
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth (Experimental): 50 patients who are randomized to the intervention group (mHealth remote monitoring devices) will be enabled with remote monitoring devices (Blood Pressure and wearable vital signs monitor, Biovotion) and "Kardia" mobile application, for home-based rehabilitation program followed by review in the outpatient Cardiology clinics.
  Interventions: Device: mHealth remote monitoring devices
- Control (No Intervention): The control group (50 patients) will just be monitored at fixed intervals in the outpatient Cardiology clinics

INTERVENTIONS:
Device: mHealth remote monitoring devices — Blood Pressure and wearable vital signs monitor, Biovotion and "Kardia" mobile application
  Arms: mHealth

SUMMARY:
This study hopes to target the remaining 80% of low risk post-myocardial infarction patients who have refused uptake the traditional cardiac rehabilitation program In Changi General Hospital. This is a 6-week home-based Cardiac rehabilitation program enabling patients to track their blood pressure, physical activity and medicine compliance through a mobile application. Each patient in the intervention arm is provided with a blood pressure monitor, activity tracker and a single lead ECG monitor. The data from these devices would be automatically synced by a mobile application and uploaded to a confidential web portal which is only accessible by physician care-givers. The application also provides educational content/tasks, appropriate reminders for taking medications and daily goals on activity targets set by the care provider. This would help to engage the patients to enable behavioural change and improve compliance to mediation and activity recommendations.

In general, 50 patients who are randomized to the intervention group (mHealth) will be enabled with remote monitoring devices (ECG, Blood Pressure, Activity tracker) and "Kardia" mobile application, for home-based rehabilitation program followed by review in the outpatient Cardiology clinics. The control group (50 subjects) will just be monitored at fixed intervals in the outpatient Cardiology clinics. Fu AT 3-4 months & 9-12 months. Subjects will be advised to commence the exercise program 2 weeks after the myocardial infarction. Block randomization using sequentially numbered sealed envelopes would be used to assign subjects to the intervention or control arms. The primary outcome measure is compliance and adherence to the "Kardia" program. Other endpoints include 6MWT, patient wellbeing and behaviour (e.g. dietary habits, stress levels, physical activity) assessed using questionnaires, major adverse cardiovascular events (MACE), modification of cardiovascular risk profiles (i.e. LDL, BP, BMI, HbA1c, etc) and medicine compliance.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the most common cause of death in Singapore, accounting for ~34% of deaths. This means 1 in every 3 deaths in Singapore is due to heart disease or stroke. Ischemic heart disease is the leading cause of mortality and accounts for 17% of all deaths attributable to life-style related risk-factors. The total burden of this disease is likely to increase given the aging population and the increase in prevalence of obesity and predisposing conditions such as diabetes mellitus, hypertension and hyperlipidaemia.

A number of modifiable environmental and patient specific factors increase the chance of developing coronary artery disease. These include smoking, high blood cholesterol, physical inactivity, diabetes, high blood pressure and obesity. Following myocardial infarction, acute coronary syndromes, surgical and percutaneous interventions, cardiac rehabilitation has provided an avenue for reducing future cardiovascular risks in patients by positively influencing these factors. The eventual goal of the program is to engage patients with permanent behavioural and life-style changes. There is strong evidence for the effectiveness of cardiac rehabilitation which is given a Class 1 recommendation from the American/European Cardiology guidelines, particularly for post-myocardial infarction patients. Several studies and meta-analyses have demonstrated a significant reduction in mortality and morbidity.

Despite the clear benefits of cardiac rehabilitation programs, the uptake of these programs has been poor due to various patient and system factors. Cardiac rehabilitation programs are traditionally carried out in hospitals and health centres under the direct personal supervision of mentoring clinicians. Patient barriers, such as time constraints and distance from treatment centres lead to poor uptake of programs among eligible patients. To overcome these barriers, home-based care models have been proposed as a viable alternative to hospital-based cardiac rehabilitation programs even in the 1980s. The current state of mobile phone communication and technology provides not only the capacity but an especially attractive media option to support home-based cardiac rehabilitation programs.

This study aims to investigate a smartphone-based cardiac rehabilitation program for patients recovering from myocardial infarction. The program focuses on providing patient centric self-monitoring platform enabling patients to take control and be actively involved in their medical care. The program ("Kardia") is a 6-week rehabilitation program enabling patients to track their blood pressure, physical activity and medicine compliance through a mobile application. Each patient in the intervention arm is provided with a blood pressure monitor and activity tracker. The data from these devices would be automatically synced by a mobile application and uploaded to a confidential web portal which is only accessible by physician care-givers. The application also provides educational content/tasks, appropriate reminders for taking medications and daily goals on activity targets set by the care provider. This would help to engage the patients to enable behavioural change and improve compliance to mediation and activity recommendations.

In Changi General Hospital, the uptake of cardiac rehabilitation among eligible patients is less than 20%. This study hopes to target the remaining 80% of patients who have refused the traditional cardiac rehabilitation program. It will be the first time that a smartphone based home cardiac rehabilitation program would be offered in Singapore. If shown to be safe and feasible, "Kardia" will help to improve patient outcomes in short to medium term. In addition, it may empower the patients to take a more active role in their medical care and promote long lasting behavioural changes in the long term. There will also be a significant operation impact if "Kardia" can be rolled out as an alternative care model to the traditional centre-based cardiac rehabilitation program, enabling greater patient access to "cardiac rehabilitation". This is also in line with national initiatives to promote an active and healthy lifestyle, i.e. National Steps Challenge by the Health Promotion Board.

The project is a randomized controlled study of smartphone based cardiac rehabilitation program compared to routine care in patients who did not sign up for traditional hospital-based cardiac rehabilitation. 50 patients who are randomized to the intervention group (mHealth) will be enabled with remote monitoring devices (Blood Pressure and wearable vital signs monitor, Biovotion) and "Kardia" mobile application, for home-based rehabilitation program followed by review in the outpatient Cardiology clinics. The control group (50 patients) will just be monitored at fixed intervals in the outpatient Cardiology clinics.

Patients will be advised to commence the exercise program 2 weeks after the myocardial infarction

Time Exercise Intensity Exercise Frequency/Duration Patient actions Week 1 light 3x/week; 10 minutes Exercise diary Week 2 light 3x/week; 20 minutes Week 3 light 3x/week; 30 minutes Week 4 moderate 3x/week; 15 minutes Week 5 moderate 3x/week; 30 minutes Week 6 moderate 4x/week; 30 minutes Week 7 moderate 5x/week; 30 minutes Week 8 moderate 5x/week; 30 minutes

ELIGIBILITY:
Inclusion Criteria:

* Age 21-85 years
* Willing and able to provide informed consent
* New onset of Post ST elevation and non-ST elevation myocardial infarction/staged PCI/acute coronary syndrome/unstable angina
* Own and able to operate App on smartphone

Exclusion Criteria:

* History of ventricular fibrillation not in the setting of acute myocardial infarction
* Documented sustained ventricular or supraventricular arrhythmia
* Unstable angina
* Awaiting staged revascularization
* Inability to perform 6MWT

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Compliance and adherence to the "Kardia" program | 9 months
  Compliance to smart phone based cardiac rehabilitation program - Uploading of completed data (BP, activity) to web portal. Compliance is defined as taking at least 1 BP per day and wearing the Biovotion for >10 hours per day.
  (90% compliance in intervention group would be considered acceptable)

SECONDARY OUTCOMES:
Improvement in 6MWT | 9 Months
  6MWT at baseline (within 2 weeks upon discharge) months 3 (+/- 2 months) and 9 (+/- 3 months) will be analysed and compared
Major Adverse Cardiovascular Events (MACE) and Hospitalizations | 12 months
  Reduction in MACE and Hospitalization
Improvement in quality of life | 9 months
  EQ5D questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Wong, MD, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dibben G, Faulkner J, Oldridge N, Rees K, Thompson DR, Zwisler AD, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2021 Nov 6;11(11):CD001800. doi: 10.1002/14651858.CD001800.pub4. PMID 34741536

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT03415841/Prot_SAP_000.pdf